CLINICAL TRIAL: NCT06947200
Title: Is There a Link Between Orthorexia Nervosa, Body Image and Psychological State in Women With Fibromyalgia Syndrome?
Brief Title: Orthorexia Nervosa in Fibromyalgia
Status: Recruiting | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH18
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- fibromyalgia group
  Interventions: Other: Fibromyalgia

INTERVENTIONS:
Other: Fibromyalgia — no intervention
  Other Names: No intervention

SUMMARY:
This clinical cross-sectional study will include 84 female patients aged between 18 and 65 years who have been diagnosed with fibromyalgia syndrome according to the 2010 American College of Rheumatology diagnostic criteria. Sociodemographic data will be recorded at the beginning of the study. Pain severity will be assessed using the Visual Analog Scale (VAS). Orthorexia nervosa-related symptoms will be evaluated with the ORTO-11 scale. Body image will be assessed with the Body Appreciation Scale 2, mood will be evaluated using the Hospital Anxiety and Depression Scale (HADS), and fibromyalgia-related impact will be assessed with the Fibromyalgia Impact Questionnaire (FIQ).

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-65 years.
* Diagnosis of fibromyalgia syndrome according to the 2010 American College of Rheumatology diagnostic criteria.
* Willingness to participate and provision of written informed consent.

Exclusion Criteria:

* Refusal to participate.
* Presence of diagnosed psychiatric disorders.
* Presence of cognitive impairment.
* Use of medications that may affect mood.

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with fibromyalgia syndrome
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
ORTO-11 Scale | Baseline
  The ORTO-11 assesses orthorexic tendencies, which refer to an unhealthy obsession with healthy eating. It consists of 11 items rated on a 4-point Likert scale. Total scores range from 11 to 44, with lower scores indicating a higher risk of orthorexia nervosa.

SECONDARY OUTCOMES:
Hospital Anxiety Scale (HADS-A): | Baseline
  The HADS-A subscale evaluates symptoms of anxiety. It consists of 7 items, each scored between 0 and 3. The total score ranges from 0 to 21, with higher scores indicating higher levels of anxiety.
Hospital Depression Scale (HADS-D): | Baseline
  The HADS-D subscale evaluates symptoms of depression. It consists of 7 items, each scored between 0 and 3. The total score ranges from 0 to 21, with higher scores indicating higher levels of depression.
Body Appreciation Scale-2 (BAS-2) | Baseline
  The BAS-2 assesses positive body image and appreciation of one's body. It consists of 10 items rated on a 5-point Likert scale (1 = Never, 5 = Always). Total scores range from 10 to 50, with higher scores indicating greater body appreciation.
Fibromyalgia Impact Questionnaire (FIQ) | Baseline
  The FIQ is a self-reported instrument designed to assess the health status and functional impact of fibromyalgia. It consists of 10 items evaluating physical functioning, work status, depression, anxiety, sleep, pain, stiffness, fatigue, and well-being. The total score ranges from 0 to 100, with higher scores indicating greater functional impairment and symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No